CLINICAL TRIAL: NCT06067672
Title: The Patient's First Point of Contact (PINPOINT) - Protocol of a Prospective Multicentre Study of Communication and Decision-making During Patient Assessments by Primary Care Practice Nurses
Brief Title: The Patient's First Point of Contact
Acronym: PINPOINT
Status: Recruiting | Type: Observational
Sponsor: University of Boras (Other)
Collaborators: Mälardalen University (Other); Netherlands Instititute for Health Services Research (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Annelie J Sundler, Professor, University of Boras
Other Study IDs: FO2023/171
Record Dates: First submitted 2023-09-25; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Nurse-Patient Relations
Keywords: Communication; Decision-making; Nurse; Primary care
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observations to investigate the current practices of communication and decision-making during Nurse-patient consultations — No intervention

SUMMARY:
The overall objective of this observational study is to investigate practices of communication and decision-making during nurses' initial assessment of patients' health problems in primary care, examine working mechanisms in good practices and develop feasible solutions.

The specific aims are:

1. To investigate patients' expectations and experiences with the communication and decision-making during their first contact with a registered nurse (RN) in primary care.
2. To investigate patient-RN communication on the level of patient involvement.
3. To investigate RNs' actual communication, assessments and decision-making, value conflicts and the challenges and strategies they use in prioritizing.
4. To analyse the underlying working mechanisms of good communication practices.
5. To develop methodologies for facilitating efficient processes in assessing, managing, and prioritizing patients in primary care for RNs.

Project PINPOINT aims for a prospective multicenter study, using various methods for data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Registered Nurses at primary care centres and patients seeking primary care for a new health concern or a new episode of a problem

Exclusion Criteria:

* Patients visiting the primary care nurse with a chronic or continuous health problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Audio-recorded observations from a purposive sample of 150 patient-nurse consultations, including 30 nurses and 150 patients will be recruited at primary care centres in three different geographic areas of the southwest of Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported expectations and experiences of the communication during consultations | At baseline (day 1), after visit (day 1) and at 2-4 weeks
  Data will be gathered with the following questionaries: QUOTE-COMM, QUality Of care Through the patients' Eyes, and The COOP/WONCA, measuring functional health status. The QUOTE-COMM is used to gather patient reported data on expectations and experiences of communication aspects during consultations. At baseline the importance of (expectations) of various communication aspects are rated, and after experiences from the consultation, to evaluate to what extent RNs met patients' expectation. The COOP/WONCA is used at baseline to measure health status.
Communication processes and patient involvement as observed during consultations | Day 1.
  Data will be gathered with audio recordings during real time consulltations. The observations with audio recordings will be coded with OPTION5, observing patient involvement in decision making, and the Verona Coding definition of emotional sequences, VR-CoDES. The OPTION5 scale is a reliable and valid instrument for investigating patient involvement in decision making. The Verona Coding Definitions on Emotional Sequences (VR-CoDES) is a reliable and valid instrument for coding of sequences of communication involving negative emotions, e.g., elicitations and expressions of patient cues and concerns, and RNs responses.

SECONDARY OUTCOMES:
Assessment and decision-making processes, and related priorities and value conflicts - from observations and RN experiences | Through study completion, an average of 1 year
  Data will be gathered with observations with audio recordings and interviews, and analysed with qualitative methods to gain insights on assessments and decision-making processes during consultations, and related priorities and value conflicts

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Sundler, Professor, Principal Investigator — University of Borås
Locations (1):
- University of Borås, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No
Data supporting these findings are not publicly available due to the participants' privacy, the General Data Protection Regulation (GDPR) law, and the ethical approval from the Swedish Ethical Review Authority.

REFERENCES:
- [Derived] Ostensson S, Acuna Mora M, Darcy L, Saarnio Huttu L, Van Dulmen S, Sundler AJ. Patient-Registered Nurse Communication: Exploring Patients' Expectations and Experience in Primary Care Consultations. Health Expect. 2025 Aug;28(4):e70353. doi: 10.1111/hex.70353. PMID 40696861
- [Derived] Sundler AJ, Heden L, Holmstrom IK, van Dulmen S, Bergman K, Ostensson S, Ostman M. The patient's first point of contact (PINPOINT) - protocol of a prospective multicenter study of communication and decision-making during patient assessments by primary care registered nurses. BMC Prim Care. 2023 Nov 29;24(1):249. doi: 10.1186/s12875-023-02208-0. PMID 38031004